CLINICAL TRIAL: NCT06199869
Title: Absence of Standard Modifiable Risk Factors Among 5000 Middle Eastern Patients With Atherosclerotic Cardiovascular Disease: Clinical Profiles and Prevalence of Other Risk Factors and Comorbidities
Brief Title: Cardiovascular Patients With no Standard Modifiable Risk Factors
Acronym: SMuRF-less-ME1
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Collaborators: The Jordan Cardiovascular Research Group JoCVRG (Other); Yarmouk University School of Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: CVA2024.SMuRFless1
Record Dates: First submitted 2023-12-25; First posted 2024-01-10 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Risk Factors
Keywords: Atherosclerotic cardiovascular disease; Standard modifiable risk factors (SMuRFs); Middle Eastern population
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of risk factors by direct interview with subjects who have atherosclerotic cardiovascular patients — Individuals identified with a diagnosis of ASCVD will fill a one page form of the associated risk factors they have

SUMMARY:
A growing number of patients develop atherosclerotic cardiovascular disease (ASCVD) despite the absence of standard modifiable risk factors (SMuRF-less). There is scarcity of studies that address this issue in the Middle Eastern population.

DETAILED DESCRIPTION:
Atherosclerotic coronary artery disease (ASCAD) claims millions of lives annually on a global level and is the leading cause of death in the Middle East. There are four standard modifiable cardiovascular risk factors (SMuRFs): hypertension, type 2 diabetes mellitus, dyslipidemia, and smoking. These are very common in the Middle East and are crucial to be screened for and addressed in an affective manner.

However, an increasing proportion of patients with ASCVD have none of these individual factors (SMuRF-less). Globally, this proportion comprises 11.6% of individuals with stable coronary disease and heart attack. No prior study has addressed the issue of the prevalence of SMuRF-less patients among the whole population of individuals with ASCVD in the Middle East.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of atherosclerotic cardiovascular disease (ASCVD).
* Ability to fill the clinical form that evaluates the presence or absence of cardiovascular risk factors including the 4 SMuRFs.

Exclusion Criteria:

* Atherosclerotic cardiovascular disease diagnosed before the age of 18 years.
* Inability to give detailed history of prespecified risk factors.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Adults (18 years of age and older) with ASCVD.
  2. ASCVD includes:
     1. Coronary heart disease
     2. stroke
     3. peripheral artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 5540 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients who do not any of the four SMuRFs | Up to 4 weeks after study enrollment
  Group of patients with definite ASCVD who do not have hypertension, diabetes, dyslipidemia or smoking.

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Istishari Hospital, Amman
  - Yarmouk University School of Medicine, Irbid

IPD SHARING:
Plan to Share IPD: Undecided
Will invite physicians to recruit 5000 individuals with ASCVD starting 1-1-2024. Once the team is gathered will share the clinical form with the all participating physicians.

REFERENCES:
- [Derived] Alrida NA, Albikawi Z, Alotaibi N, Alkouri O, Saifan AR, Jarrah M, Hammoudeh A, Khader Y, Alenezy A, Al-Zu'bi BM, Alharbi A, Alhalaiqa F, AbuRuz ME. Association of SMuRFs with cardiovascular risk factors, disease burden, and pharmacological management in Middle Eastern patients with ASCVD and a family history of premature CVD. Front Cardiovasc Med. 2025 Nov 27;12:1678767. doi: 10.3389/fcvm.2025.1678767. eCollection 2025. PMID 41393265
- [Derived] Alkouri O, Alrida NA, Alabkal RM, Khader Y, Albikawi Z, Ababneh A, Alobaidly A, Qaladi O, Alharbi A, Jarrah M, Alotaibi N, Al-Bashaireh AM, Hammoudeh A, AbuRuz ME, Almustafa LA, Khraisat O, Al-Nsair N. Prevalence of physical activity and its association with atherosclerotic cardiovascular risk factors in young women in the middle east: a sub-analysis of the ANCHORS study. BMC Public Health. 2025 Oct 1;25(1):3268. doi: 10.1186/s12889-025-24595-y. PMID 41034877
- [Derived] Hammoudeh AJ, Aldalal'ah M, Smadi EA, Alrishoud D, Alomari A, Alkhawaldeh M, Rizik A, Okour MF, Araydah M. Absence of Standard Modifiable Risk Factors in Middle Eastern Patients with Atherosclerotic Cardiovascular Disease. The Jordan Absence of Standard Modifiable Risk Factors (SMuRF-Less) Study. Vasc Health Risk Manag. 2025 Feb 5;21:39-50. doi: 10.2147/VHRM.S499355. eCollection 2025. PMID 39931041